CLINICAL TRIAL: NCT04045353
Title: A Randomized Trial of a Low Carbohydrate Diet Versus the Current Recommended Dietary Guidelines to Improve Health Outcomes in Obese Postpartum Women
Brief Title: A Study of a Low-Carbohydrate Diet to Improve Maternal Health After Childbirth
Acronym: SLIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0314
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Postpartum Weight Retention; Insulin Sensitivity
Keywords: Low carbohydrate diet
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (No Intervention): Subjects will receive standard counseling on obesity as part of routine postpartum care.
- Low carbohydrate diet education (Active Comparator): Subjects will receive educational materials regarding a low carbohydrate diet in addition to the standard counseling on obesity as part of routine postpartum care.
  Interventions: Behavioral: Low carbohydrate diet education
- Low carbohydrate diet education with behavioral component (Active Comparator): Subjects will receive in person instruction regarding a low carbohydrate diet as part of a 12 week course, in addition to receiving educational materials regarding a low carbohydrate diet and the standard counseling on obesity as part of routine postpartum care.
  Interventions: Behavioral: Low carbohydrate diet education; Behavioral: Low carbohydrate diet education with behavioral component

INTERVENTIONS:
Behavioral: Low carbohydrate diet education — A 200 page informational document that connects with an online application will be provided to subjects.
  Arms: Low carbohydrate diet education; Low carbohydrate diet education with behavioral component
Behavioral: Low carbohydrate diet education with behavioral component — A 12 week course taught be a certified instructor will teach subjects about a low carbohydrate document. Subjects will also be given a 200 page informational document that connects with an online application.
  Arms: Low carbohydrate diet education with behavioral component

SUMMARY:
The study is evaluating the effects of a standard diet to a low carbohydrate diet in obese women after having a baby. The purpose of the study is to determine if a low carbohydrate diet is associated with improvement in insulin sensitivity in postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at University of Texas Medical Branch
* Body max index greater than or equal to 30 kilograms/meters squared at the final prenatal visit prior to delivery.
* Singleton gestation.
* Accessibility to the internet.
* Basic understanding and comprehension of the English language to be assessed by study personnel at the time of recruitment.

Exclusion Criteria:

* Diabetes mellitus on medication.
* Serious medical condition, such as heart failure, kidney failure, or severe asthma, as determined by the principle investigator.
* Planned pregnancy during study period.
* Enrolled in another trial that may affect outcome.
* Subject unlikely to be followed up after delivery.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is limited subjects that are postpartum; therefore, can only include female participants.
Enrollment: 11 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity as measured by homeostatic model assessment of insulin sensitivity. | Baseline, 3 months
  Homeostatic model assessment for measurement of insulin sensitivity will be computed with fasting insulin and glucose levels (fasting for at least 8 hours) with the following calculation: (glucose x insulin/22.5). This calculation is measured in molar units (mmol/L).

SECONDARY OUTCOMES:
Change in insulin sensitivity as measured by homeostatic model assessment of insulin sensitivity. | Baseline, 6 months
  Homeostatic model assessment for measurement of insulin sensitivity will be computed with fasting insulin and glucose levels (fasting for at least 8 hours) with the following calculation: (glucose x insulin/22.5). This calculation is measured in molar units (mmol/L).
Change in weight measured in pounds. | Baseline, 3 months
  The subject will be weighed at baseline and at 3 months.The weight will be calculated in pounds.
Change in weight measured in pounds. | Baseline, 6 months
  The subject will be weighed at baseline and at 6 months. The weight will be calculated in pounds.
Development of diabetes postpartum as measured by 2 hour glucose tolerance test. | 3 months
  As part of routine postpartum care, women at risk for diabetes have a glucose tolerance test performed within 3 months postpartum.
Change in blood pressure as measured by blood pressure cuff in mmHg. | Baseline, 3 months
  The subject will have blood pressure checked at baseline and at 3 months. Blood pressure will be calculated in mmHg.
Change in blood pressure as measured by blood pressure cuff in mmHg. | Baseline, 6 months
  The subject will have blood pressure checked at baseline and at 6 months. Blood pressure will be calculated in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Sara O Jacobs, MD, Principal Investigator — University of Texas; Antonio Saad, MD, Principal Investigator — University of Texas; Ashley Salazar, WHNP, Study Director — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morkrid K, Jenum AK, Sletner L, Vardal MH, Waage CW, Nakstad B, Vangen S, Birkeland KI. Failure to increase insulin secretory capacity during pregnancy-induced insulin resistance is associated with ethnicity and gestational diabetes. Eur J Endocrinol. 2012 Oct;167(4):579-88. doi: 10.1530/EJE-12-0452. Epub 2012 Aug 13. PMID 22889687
- [Background] Rooney BL, Schauberger CW. Excess pregnancy weight gain and long-term obesity: one decade later. Obstet Gynecol. 2002 Aug;100(2):245-52. doi: 10.1016/s0029-7844(02)02125-7. PMID 12151145
- [Background] Foster GD, Wyatt HR, Hill JO, McGuckin BG, Brill C, Mohammed BS, Szapary PO, Rader DJ, Edman JS, Klein S. A randomized trial of a low-carbohydrate diet for obesity. N Engl J Med. 2003 May 22;348(21):2082-90. doi: 10.1056/NEJMoa022207. PMID 12761365

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT04045353/Prot_SAP_001.pdf